CLINICAL TRIAL: NCT02913495
Title: Vaginal Versus Intramuscular Progesterone for the Prevention of Recurrent Preterm Birth
Acronym: VIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Baystate Medical Center (Other); George Washington University (Other); Vriginia Commonwealth University (Unknown); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16D.542
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Premature Birth
Keywords: Progesterone; Prevention of preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Progesterone (Experimental): 200mg micronized progesterone vaginally, to be taken daily starting at 16 0/7 - 23 6/7 weeks, and continued daily until 36 6/7 weeks' gestation or delivery
  Interventions: Drug: Vaginal Progesterone
- Intramuscular Progesterone (Active Comparator): 250mg intramuscular progesterone to be administered weekly starting at 16 0/7 - 23 6/7 weeks, and continued weekly until 36 6/7 weeks' or delivery.
  Interventions: Drug: Intramuscular Progesterone (17 alpha hydroxprogesterone caproate)

INTERVENTIONS:
Drug: Vaginal Progesterone
  Other Names: micronized progesterone
  Arms: Vaginal Progesterone
Drug: Intramuscular Progesterone (17 alpha hydroxprogesterone caproate)
  Other Names: Makena
  Arms: Intramuscular Progesterone

SUMMARY:
The purpose of this study is to evaluate the two suggested therapies for prevention of recurrent preterm birth (PTB) in women with a prior spontaneous preterm birth, vaginal and intramuscular progesterone to determine whether vaginal progesterone is superior to intramuscular progesterone in the prevention of recurrent preterm birth.

DETAILED DESCRIPTION:
Preterm birth is one of the leading causes of neonatal morbidity and mortality. One of the greatest predictors of preterm birth is a history of prior spontaneous preterm birth. Presently 17 hydroxyprogesterone caproate (intramuscular) is the only FDA approved product for the prevention of recurrent preterm birth, however recent studies suggest that vaginal progesterone may be used for this purpose, and may even be superior. The American College of Obstetrics and Gynecology does not specify the optimal route of progesterone administration for the prevention of recurrent preterm birth. It is our intention to compare vaginal and intramuscular progesterone to see if one is superior.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies
* ≥18 years old
* Estimated gestational age less than 24 0/7 weeks
* Prior spontaneous preterm birth of a singleton pregnancy between 16 0/7-36 6/7 weeks.
* Patients are also required provide consent, demonstrate an understanding of the purpose of the study, and agree to the study protocol.

Exclusion Criteria:

* History of an adverse reaction to progesterone;
* A contraindication to progesterone treatment;
* Placenta previa or accreta;
* Major fetal anomaly diagnosed on ultrasound or known chromosomal disorder;
* Multifetal gestation;
* Preterm labor, premature rupture of membranes, or clinical chorioamnionitis, at the time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Preterm birth <37 weeks | up to 9 months (delivery)
  Incidence of gestational age of delivery less than 37 weeks

SECONDARY OUTCOMES:
Gestational age of delivery | up to 9 months (delivery)
Preterm birth <34 weeks and <28 weeks | up to 9 months (delivery)
Second trimester cervical length <25mm | 2 months
Mode of delivery | up to 9 months (delivery)
  Delivery mode- vaginal, cesarean, operative vaginal
Maternal mortality | up to 9 months (delivery)
5 minute Apgar score | up to 9 months (delivery)
Neonatal intensive care unit admission | up to 9 months (delivery)
Composite neonatal morbidity | up to 9 months (delivery)
  (respiratory distress syndrome, grade III or IV intraventricular hemorrhage, culture proven sepsis, neonatal enterocolitis, and perinatal mortality up to 28 days of life)
Birthweight | up to 9 months (delivery)
Perinatal mortality up to 28 days of life | up to 10 months (4 weeks after delivery)
Medication side effects | up to 9 months (delivery)
Satisfaction with medication (5 point Likert scale) | up to 9 months (delivery)
Medication adherence | up to 9 months (delivery)
  Vaginal progesterone:
  * Overall adherence: #days used/#days of treatment x 100
  * Non-adherent: ≥4 days between doses
  Intramuscular progesterone:
  * Overall adherence: #weeks used/#weeks of treatment x 100
  * Non-adherent: ≥10 days between doses
Planned subgroup analysis for the outcome preterm birth <37 weeks, <34 weeks, <28 weeks | up to 9 months (delivery)
  Planned subgroup analysis for the primary outcome as well as the secondary outcomes of preterm birth <34 weeks and <28 weeks of patients with a cervical length <25mm versus ≥25mm, history-indicated cerclage versus not, and for those started on progesterone 16-20 weeks versus 20-24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rupsa C Boelig, MD, Principal Investigator — Thomas Jefferson University Hospital; Sidney Kimmel Medical College
Locations (3):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Baystate Medical Center, Springfield, Massachusetts
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Results will be available, individual participant data may not be

REFERENCES:
- [Background] Committee on Practice Bulletins-Obstetrics, The American College of Obstetricians and Gynecologists. Practice bulletin no. 130: prediction and prevention of preterm birth. Obstet Gynecol. 2012 Oct;120(4):964-73. doi: 10.1097/AOG.0b013e3182723b1b. No abstract available. PMID 22996126
- [Background] Saccone G, Khalifeh A, Elimian A, Bahrami E, Chaman-Ara K, Bahrami MA, Berghella V. Vaginal progesterone vs intramuscular 17alpha-hydroxyprogesterone caproate for prevention of recurrent spontaneous preterm birth in singleton gestations: systematic review and meta-analysis of randomized controlled trials. Ultrasound Obstet Gynecol. 2017 Mar;49(3):315-321. doi: 10.1002/uog.17245. Epub 2017 Feb 6. PMID 27546354
- [Derived] Boelig RC, Schoen CN, Frey H, Gimovsky AC, Springel E, Backley S, Berghella V. Vaginal progesterone vs intramuscular 17-hydroxyprogesterone caproate for prevention of recurrent preterm birth: a randomized controlled trial. Am J Obstet Gynecol. 2022 May;226(5):722.e1-722.e12. doi: 10.1016/j.ajog.2022.02.012. Epub 2022 Feb 19. PMID 35189093